Narcotic-Free Percutaneous Nephrolithotomy NCT05924165 PI: Mantu Gupta, MD Document Date: 4-9-2024

## 

Study ID: STUDY-23-00206 Form Version Date: 04May2023

#### STUDY INFORMATION:

Study Title: Narcotic-Free Percutaneous Nephrolithotomy

Study site(s): Mount Sinai West

Principal Investigator (Lead Researcher): Mantu Gupta, MD

**Physical Address:** 425 W. 59<sup>th</sup> Street, Suite 4F. New York, NY 10019 **Mailing Address:** 425 W. 59<sup>th</sup> Street, Suite 4F. New York, NY 10019

**Phone:** 212-241-1272

### **SUMMARY OF THIS RESEARCH STUDY:**

This document explains a research study you might be interested in joining. Participation in the study is voluntary. You can agree to join or not. Your decision will not limit your ability to receive care at Mount Sinai. You should only agree to take part if you understand the study and if all of your questions about the research study are answered. If you do join the study, the research team must share any new information with you that may change your mind about taking part.

The purpose of this research study is to determine if a non-steroidal anti-inflammatory drug (NSAID) called ketorolac (similar to ibuprofen) is an effective alternative to narcotic pain medication (oxycodone) following kidney stone removal surgery (percutaneous nephrolithotomy).

If you choose to take part, no additional visits are required, and there is only a minimal change from the normal standard of care. You will be asked to:

- Complete a brief, one question survey regarding your pain levels via telephone call for the first five days after surgery.
- Bring your leftover medication that was prescribed to you after surgery to your follow up appointment for a pill count
- Complete a five-minute survey during your follow up appointment regarding your pain/discomfort and post operative experience
- Agree to have private information study data stored for the duration of the study. Once the study is complete, your data will be de-identified.
- There is no payment for taking part in the study.

If you choose to take part, the main risks to you are potential side effects from each medication. The main risks associated with ketorolac include gastrointestinal upset and renal impairment (although this

-----FOR IRB USE ONLY------

Rev 11.11.2022



### 


is very rare). The main risks associated with oxycodone include constipation and nausea/vomiting. A full list of potential side effects can be found in the risks section of this consent form. If you run out of medication, your pain is not well controlled, or if you are having side effects from your medication, please call our 24-hour phone number (212-241-1272) to speak to a member of our team. Our team will prescribe you additional medication or a different medication to help with your pain.

You will not benefit directly from taking part in this research.

Instead of taking part in this research, you may have your kidney stone removal surgery without taking part in this research study. As part of standard care your physician may prescribe either ketorolac, oxycodone or some other pain medication for postoperative pain management.

If you are interested in learning more about this study, please continue to read below.

#### STUDY PARTICIPATION:

You may qualify to take part in this research study because you are scheduled to undergo kidney stone removal surgery, called percutaneous nephrolithotomy (PCNL).

Your participation in this research study is expected to last 10-14 days.

There are 90 people expected to take part in this research study at Mount Sinai West.

Funds for conducting this research study are provided by Mount Sinai.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### **DESCRIPTION OF WHAT IS INVOLVED:**

If you agree to take part in this research study, here is what may be involved:

- o On the day of surgery, you will undergo PCNL with your study doctor according to the standard of care
- o Following surgery, you will be randomly assigned to one of two groups which will decide what medications are prescribed to you for postoperative pain:
  - 1. Ketorolac (an NSAID medication similar to ibuprofen)
  - 2. Oxycodone (a narcotic medication)

Rev 11.11.2022



## 


- o Both medications are routinely prescribed after PCNL and considered normal standard of care.
- Following surgery, a member of the research team will ask you what your pain level is on a scale of 1-10.
- For the first ten days after surgery, a member of the research team will follow up with you via telephone call to ask you what your pain level is on a scale of 1-10 (for the first five days) and if you are experiencing any side effects (for all ten days).
- When you return to the office for your stent removal 10-14 days after surgery, you will be instructed to bring back all your unused medication so that we can conduct a pill count. A team member will call you 24 hours before your appointment for an additional reminder.
- At your follow up appointment, you will be asked to complete a five-minute survey about your postoperative pain and experience. You will also be asked to rate your pain on a scale of 1-10.
- o After the surveys and pill count are done, your participation in the study is complete.

### Randomization

No one, not you, or anyone from your medical team or from the research team will be able to choose what post operative medication you are prescribed. It will be by chance, like flipping a coin. You will have an equal one in two chance of being given each medication.

## **Pregnancy**

If you can possibly get pregnant, a urine test for pregnancy will be done before you begin the study on the day of surgery.

You cannot be included in the study if you are or become pregnant, as the study drugs could harm your fetus. You also should not be in the study if you are producing milk to feed a child as the study drug could harm your baby.

Unless you are at least one year past menopause or have had a successful operation to make pregnancy impossible, you should use at least two methods of effective birth control. Unless you are sexually abstinent (not having genital sex) the recommended methods of birth control are:

- The consistent use of approved hormonal birth control (pill, patches, or rings),
- An intrauterine device (IUD),
- Contraceptive injection (Depo-Provera),
- Double barrier methods (Diaphragm with spermicidal gel or condoms with contraceptive foam),
- Sexual abstinence (no sexual activity),
- Sterilization (a vasectomy, getting tubes tied, or a hysterectomy).

All birth control methods (other than abstinence and sterilization) are only effective if you use them properly, start them at least one month before you begin the research study, and continue using them throughout the research study and for one month after the research study ends. If you are unsure

Rev 11.11.2022



## 


whether the method of birth control you use is approved to use while you are in this study, you should ask the Lead Researcher before you begin the study. If you are less than one-year post-menopausal, you could still become pregnant. If you or your partner becomes pregnant, or may be pregnant, at any time during the study, you must tell a person from the research team immediately. The team may stop the study drug and refer you/your partner to an obstetrician/gynecologist for follow-up.

Should you/your partner become pregnant, whether or not you/your partner have the baby, the people funding and overseeing the research may ask for information on the pregnancy, even if you are no longer part of the study. You/your partner will be asked for additional written consent to share this information if that happens.

## **USE OF YOUR DATA AND/OR SAMPLES:**

In addition to being used to complete this research study, your personal information (such as, name, address, date of birth, social security number), and study data may also be used and shared for additional (future) research. Before anything is shared, all of your identifying personal information will be removed and it will be replaced with a code. Researchers are not planning on giving you the details of any of this future research nor the results. That means that a research project might be done that you would not consent to if provided with the details of that research project. If you do not want any future research to be done with your data, even with your identity removed, please do not sign this consent form or take part in the study.

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study, you will be responsible for the following things:

- Follow the directions of the study doctor and study staff.
- Allow us to follow your care for 10-14 days and access your medical records
- Complete the telephone survey for the first five days after surgery
- Return to the office for your follow up appointment and take the five minute survey given to you.
- Call our 24-hour phone number (212-241-1272) if you run out of medication, are experiencing severe pain, or you are experiencing side effects from your medication.

## COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

You will not be paid for taking part in this study. Being in this study will not cost you anything extra.

#### **POSSIBLE BENEFITS:**

This study is not designed to benefit you personally. However, we hope the information from this study will provide valuable data on the pain medications needed after kidney stone surgery.

Rev 11.11.2022



## 


### **POSSIBLE RISKS AND DISCOMFORTS:**

- Physical risks include side effects for each medication:
  - Risks associated with oxycodone include constipation, nausea, vomiting, headache, pruritus (itchy skin), insomnia (trouble sleeping), dizziness, asthenia (weakness/tiredness), and somnolence (drowsiness).
  - Risks associated with ketorolac include:
    - Gastrointestinal and bleeding risks: nausea, vomiting, diarrhea, gas, peptic ulcers, gastrointestinal bleeding, and/or perforation of the stomach or intestines
    - Cardiovascular risks: serious cardiovascular thrombotic events (blood clots), myocardial infarction (heart attack), stroke, hypertension
    - Renal (kidney) risks: renal impairment (this is rare because your baseline renal function is normal).
    - Other risks: dizziness, drowsiness, mental/mood changes, allergic reactions (rare)
- Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.
- Group Risks Although your name will not be given to researchers, basic information such
  as your race, ethnic group, and sex may be shared. This information helps researchers
  learn whether the factors that lead to health problems are the same in different groups of
  people. It is possible that such findings could one day help people of the same race, ethnic
  group, or sex as you. However, they could also be used to support harmful stereotypes or
  discrimination.
- Privacy Risks Your name and other information that could directly identify you (such as an address, date of birth, or social security number) will never be placed into a database. However, because your genetic information is unique to you, there is a small chance that someone could trace it back to you. The risk of this happening is very small, but may grow in the future. Since the database contains genetic information, a break in security may also pose a potential risk to blood relatives as well as yourself. For example, it could be used to make it harder for you (or a relative) to get or keep a job or insurance. If your private information was misused, it is possible you would experience other harms, such as stress, anxiety, stigmatization, or embarrassment from revealing information about your family relationships, ethnic heritage, or health conditions.

#### OTHER OPTIONS TO CONSIDER:

You may decide not to take part in this research study. If you decide not to take part, this will not affect the clinical care you receive at Mount Sinai. The choice is totally up to you.

-----FOR IRB USE ONLY------

Rev 11.11.2022



### 


Instead of being in this research study, you can still have the kidney stone removal surgery described in this study.

### IN CASE OF INJURY DURING THIS RESEARCH STUDY

If you are injured or made sick from taking part in this research study, you will get medical care. Generally, it will be billed to you or your insurance. You will be responsible for all treatment costs not covered by your insurance, including deductibles, copayments, and coinsurance. This does not prevent you from seeking payment for injury related to malpractice or negligence. You can contact the Lead Researcher for more information.

#### **ENDING PARTICIPATION IN THE RESEARCH STUDY:**

You may stop taking part in this study at any time. No matter what you choose, your care and benefits through Mount Sinai will not be negatively impacted.

If you decide to stop being in the study, please contact the Lead Researcher or the research staff.

You may also withdraw your permission for the researchers to use and share any of your protected information for research, but <u>you must do so in writing</u> to the Lead Researcher at the address on the first page. Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected if that information is necessary to complete the research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

If you decide you don't want your data to be used for research anymore, you can contact the researcher and ask to have your data withdrawn or labeled so that they will not to be used in additional projects or shared. If your data have already been shared with researchers, those researchers will be asked to stop using them. However, if any data has already been shared without your identity or a linking code, it won't be possible to retrieve them. Data that have already been used will not be affected by your decision. If your data have already been deposited in an external repository, the study team will request that your data be removed.

<u>Withdrawal without your consent</u>: The Lead Researcher, the funder or Mount Sinai may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the research team have not been followed, the Lead Researcher believes it is in your best interest, or for any other reason. If data have been stored as part of the research study, they too can be destroyed without your consent.

-----FOR IRB USE ONLY------

Rev 11.11.2022



### 

| Study ID | : STUE | )Y- <b>23</b> - | 00206 |
|--------------|--------|-----------------|-------|
| Form Versior | Date: | 04Ma | y2023 |

#### **CONTACT INFORMATION:**

If you have any questions, concerns or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Lead Researcher at phone number 212-241-1272.

### **DISCLOSURE OF FINANCIAL INTERESTS:**

Researchers sometimes get paid for consulting or doing work for companies that produce drugs, biologics or medical devices. If you have questions regarding industry relationships, you are encouraged to talk to the Lead Researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

#### **MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:**

As part of this study, some of your private and/or protected health information will be obtained, used, and shared with your permission. There is a Federal Health Insurance Portability and Accountability Act (HIPAA) that makes sure this is done correctly and safely.

### What is protected health information (PHI)?

PHI is the combination of two things:

- 1. PHI contains information that identifies you. It will be used to contact you and link you to your health information, like name, date of birth, medical record number, and address.
- 2. PHI also contains health information, including information about your mental and physical health from your visits to doctors or hospitals, or from study visits.

Every time you visit a hospital or your doctor, PHI is created and recorded in your medical record by your healthcare providers. In the same way, the PHI created as part of this study will be linked to who you are and your medical information.

What PHI is collected and used in this research study, and might also be shared with others?

As part of this study, the research team at the hospital(s) involved in the research will collect your address, telephone number, dates directly related to you (birth, admission, discharge, follow up date), and medical records number.



## 


During the study, the researchers will gather information by:

- Reviewing and/or taking your medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- Doing a physical examination that generally also includes blood pressure reading, heart rate, breathing rate, and temperature.
- Completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.

### Why is your PHI being used?

Researchers need the information that identifies you so they can contact you during the study. They need your health information and the results of any tests and procedures being collected as part of this study to answer the questions posed in the study. The purpose of the study is discussed earlier in this consent form. Before researchers analyze the data, they remove any information that would let others know who you are or that you took part in the study. If researchers publish or present study results at scientific meetings, lectures, or other events, their presentations would not include any information that would let others know who you are, unless you give separate permission to do so.

The Lead Researcher may also use and share the results of these tests and procedures with other healthcare providers at Mount Sinai who are involved in your care or treatment. The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example:

- The Mount Sinai Program for the Protection of Human Subjects is responsible for overseeing research on human participants and may need to see your information.
- If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes.
- If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

#### Who, outside Mount Sinai, might receive your PHI?

As part of the study, the Lead Researcher, research team and others in the Mount Sinai workforce may disclose your PHI, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Lead Researcher.)

- The United States Department of Health and Human Services (DHHS) and the Office of Human Research Protection (OHRP) (the government organization that is responsible for protecting human research participants).

In all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier unless disclosure of the direct

Rev 11.11.2022



## 


identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Lead Researcher will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board (IRB) allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, OHRP, as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

### For how long will Mount Sinai be able to use or disclose your PHI?

Your authorization for use of your PHI for this specific study does not expire.

### Will you be able to access your records?

During your participation in this study, you will have access to your medical record and any study information that is part of that record. The research team is not required to release research information to you that is not part of your medical record.

### Do you need to give the researchers permission to obtain, use or share your PHI?

NO! If you decide not to let the research team obtain, use or share your PHI, you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment, or enrollment in any health plans or affect your eligibility for benefits.

### Can you change your mind?

If you decide to stop being in the study, please contact the Lead Researcher or the research staff. The research team may ask you whether they can continue to collect information from your medical record. You will also have to decide if you wish to limit the continued use of the information collected during the study. Under US privacy laws you may also withdraw your permission for the researchers to use and share any of your protected information for research, but you must do so in writing to the Lead Researcher at the address on the first page.

Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected, but only to complete this research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

------FOR IRB USE ONLY------



Effective Date: 4/9/2024 End Date:4/8/2025

Rev 11.11.2022

## 


It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If researchers are reviewing your medical records or asking questions about your medical history or conditions, it is possible that they may learn information related to your HIV status. If that is the case, the following information concerns you. If researchers are not reviewing your medical records or asking questions about your medical history or conditions, then you may ignore the following section.

## **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 306-5070. These agencies are responsible for protecting your rights.

## How the Institutional Review Board (IRB) can help you:

This research has been reviewed and approved by an Institutional Review Board (IRB). You may reach a representative of the Mount Sinai Program for Protection of Human Subjects at telephone number (212) 824-8200 during regular work hours (Monday-Friday, 9am-5pm, excluding holidays) for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

| FOR IRB USE ONLY |
|------------------|



Rev 11.11.2022

## 


| Printed Name of Participant | Date | Time |
|---|---|---|
| AND OBTAINING CONSENT: | | |
| Printed Name of Consent Delegat | e Date | Time |
| lained to, and apparently understoo | | - |
| Printed Name of Witness | Date | Time |
| | AND OBTAINING CONSENT: Printed Name of Consent Delegate that the information in the consent delained to, and apparently understood participant. | AND OBTAINING CONSENT: Printed Name of Consent Delegate Date that the information in the consent document and plained to, and apparently understood by, the paraparticipant. |

